CLINICAL TRIAL: NCT06078696
Title: Siplizumab-based Conditioning for Hematopoietic Stem Cell Transplantation in Patients With Advanced Sickle Cell Disease (CD2 SCD)
Brief Title: Siplizumab for Sickle Cell Disease Transplant
Acronym: CD2 SCD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: ITB-Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAU5053
Record Dates: First submitted 2023-08-30; First posted 2023-10-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Anemia, Sickle Cell
Keywords: hemoglobin S (HbS) Disease; Hemoglobin S Disease; Sickle Cell Disease; Sickle Cell Disorders; Sickling Disorder Due to Hemoglobin S; Advanced Sickle Cell Disease; Sβ0 thalassemia; Advanced SCD
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait; Disease | interventions — siplizumab; Exchange Transfusion, Whole Blood; Whole-Body Irradiation; Cyclophosphamide; Mesna; Sirolimus; Rituximab; Biosimilar Pharmaceuticals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Siplizumab (Experimental): Participants will receive 5 infusions of siplizumab. The first dose is given 14 days prior to the infusion of stem cells; the second dose is given 6 days before infusion; and doses 3, 4, and 5 are given on the day before, day of, and day after stem cell infusion.
  Interventions: Drug: Siplizumab; Procedure: Exchange Transfusion; Procedure: Total Body Irradiation; Procedure: Stem Cell Infusion; Drug: Cyclophosphamide 50mg; Drug: Mesna; Drug: Sirolimus Oral Tablet; Drug: Rituximab or Biosimilar

INTERVENTIONS:
Drug: Siplizumab — Premedication with diphenhydramine 50 mg PO is to be given 1 hour prior to siplizumab infusion. Premedication with hydrocortisone succinate 100 mg IV infused over 30 minutes and acetaminophen 650 mg PO are to be given at least 30 minutes prior to siplizumab infusion. Siplizumab 4.8 mg/kg total is given on Day -14 and 0.6mg/kg is given on days -6, -1, 0, and +1. It will be given as an IV infusion over 1 hour.
  Other Names: TCD601 (Siplizumab)
Procedure: Exchange Transfusion — Patient will undergo a red blood cell exchange transfusion to achieve a Hemoglobin S (HgbS) level < 20% prior to starting therapy to prevent the development of a vaso-occlusive Crisis (VOC).
Procedure: Total Body Irradiation — Radiation dose is 2Gy (Gy is a radiation unit of measurement). Radiation source and dose rates will be according to institutional practice. Total Body Irradiation (TBI) may be delivered from either linear accelerator or Cobalt sources.
  Other Names: TBI
Procedure: Stem Cell Infusion — Standard institutional procedures should be followed for the processing and administration of stem cell products for infusion. The infused graft under no circumstances is to be irradiated. No in-line leukocyte filter should be used and no medications or fluids should be given piggyback through the catheter lumen used for infusion of stem cells. Vital signs should be monitored before beginning the infusion and periodically during administration and in accordance with institutional guidelines. Pre-medications prior to the graft infusion will be according to the institutions standard practice. Benadryl, epinephrine, hydrocortisone, and oxygen be available at the bedside, as well as an emergency medical code cart available in the vicinity of the patient, for emergency use in case of an infusion reaction.
Drug: Cyclophosphamide 50mg — Cyclophosphamide will be given on days +3 and +4 at a dose of 50 mg/kg. Hydration prior to cyclophosphamide should be given according to standard institutional practice. Day +3 dose should occur between 60 and 72 hours after graft infusion and day +4 post-transplant should occur approximately 24 hours after prior dose. Cyclophosphamide will be given as an IV infusion over 1-2 hours depending on volume or as per institutional standard practice. Cyclophosphamide will be dosed according to adjusted ideal body weight (AIBW) in patients weighing > 125% ideal body weight (IBW).
  Other Names: Cytoxan; Cytoxan Lyophilized
Drug: Mesna — Mesna is to be given starting 1 hour prior to cyclophosphamide at the same dose (50 mg/kg) as a continuous infusion over 24 hours.
  Other Names: Mesnex
Drug: Sirolimus Oral Tablet — Sirolimus will be given orally with a loading dose of 12 mg, then followed by 4 mg orally daily. Dosage will be adjusted to a therapeutic target of 10 - 15ng/ml in first 3 months post transplant and 3-10 after 3 months. Sirolimus should be started on day +5. It will be continued until at least day 180. Sirolimus can be tapered or continued according to the treating physician discretion and the presence of absence of GVHD and/or degree of donor chimerism. Sirolimus should be continued if donor chimerism is less than 50% to prevent graft loss.
  Other Names: Rapamycin; Rapamune
Drug: Rituximab or Biosimilar — Rituximab (375 mg/m2/dose) will be administered on Days -14 and -6. In those subjects receiving ongoing renal replacement therapy, rituximab should be administered several hours after hemodialysis. The first rituximab solution for infusion should be administered intravenously at an initial rate of 50 milligrams/hour (mg/hr). The rate may be escalated by 50mg/hr every 30 minutes to a maximum of 400 mg/hr. Subsequent infusions may be started at 100 milligrams/hour (mg/hr) and titrated by 100 mg/hr every 30 minutes to a maximum of 400mg/hr if the subject tolerated the first infusion.
  Other Names: Riabni; Rituxan; Ruxience; Truxima

SUMMARY:
The purpose of this study is to find out whether siplizumab is safe and effective for patients with SCD undergoing an allogeneic transplant and to prevent development of Graft versus Host Disease (GVHD) and graft failure. The main goals of this study are :

* To determine if acute GVHD occurs and how severe the acute GVHD is in subjects receiving the study drug
* To determine if graft failure occurs in subjects receiving the study drugs

In this study, participants will receive 5 infusions of the study drug, siplizumab, while getting a stem cell transplant for SCD. Before siplizumab infusion, participants will be given medications to reduce the risks of allergic reaction to the drug.

DETAILED DESCRIPTION:
Phase I/II label single arm safety assessment study of Siplizumab-based conditioning. It is designed to determine the safety and feasibility of hematopoietic stem cell transplantation for patients with advanced sickle cell disease using in vivo T cell depletion with Siplizumab.

It is a three-stage design with a target sample size of at most 18 patients. At the first stage, a total of 6 patients will be recruited, the study will be stopped, if 2 or more of patients experience any of the following events: graft failure/Grade 3-4 acute GVHD/death in the first 100 days. If not, the study will proceed to the second stage and recruit additional 6 patients. The study will be stopped if 4 or more patients experience an event as specified above among the 12 patients. If not, the study will proceed to the third stage and recruit additional 6 patients, the study will be stopped any time if 6 or more patients experience an event among the 18 patients. The study will be stopped at any time if a patient death occurs.

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Patients with sickle cell anemia (Hb SS, Sβ0 thalassemia or severe SC) who are 18 - 50 years of age inclusive AND who have 1 or more of the following:

   1. Clinically significant neurologic event (stroke) or any neurological deficit lasting at least 24 hours. Stroke will be defined as a clinically significant neurologic event that is accompanied by an infarct on cerebral MRI or cerebral arteriopathy requiring chronic transfusion therapy.
   2. History of two or more episodes of ACS in the 2-year period preceding enrollment despite supportive care measures (i.e. asthma therapy and/or hydroxyurea).
   3. History of three or more severe vaso-occlusive pain crises per year in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea).
   4. Administration of regular red blood cell (RBC) transfusion therapy, defined as receiving 8 or more transfusions per year for 1 year or more to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and ACS)
   5. An echocardiographic finding of tricuspid valve regurgitant jet (TRJ) velocity > or equal to 2.7 m/sec or pulmonary hypertension diagnosed by right heart catheterization.
   6. Chronic kidney disease including patients on hemo-dialysis
   7. Recurrent tricorporal priapism defined as at least 2 episodes of an erection last ≥4 hours involving the corpus cavernosa and corpus spongiosa.
   8. Recipient cannot be pregnant or lactating.
2. Adequate organ functions as defined as:

   1. Eastern Cooperative Group (ECOG) performance status of 2 or better
   2. Cardiac function: left ventricular ejection fraction (LVEF) of 40% or greater
   3. Pulmonary Function: Pulse oximetry with a baseline oxygen saturation of 85% or greater and corrected diffusing capacity of the Lungs for carbon monoxide (DLCO) of 35% or greater
   4. Hepatic Function: Serum conjugated (direct) bilirubin less than 3x upper limit of normal for age as per local laboratory, alanine aminotransferase (ALT) and aspartate transaminase (AST) less than 5 x upper limit of normal as per local laboratory. Patients whose hyperbilirubinemia is the result of hyperhaemolysis, or a sever drop in hemoglobin post blood transfusion are not excluded.
   5. Absence of liver cirrhosis, bridging fibrosis and active hepatitis as documented by liver biopsy for patients with evidence of iron overload by serum ferritin or MRI. The histological grading and scale described by Ishak and colleagues (1995) will be used.
3. Patient must have a matched-or mismatched unrelated donor or mismatched related family donor.

   1. For HLA-matching we will assess 12 HLA-antigens (HLA-A, B, C, DRB1, DQB1 and DPB1).
   2. Fully matched unrelated transplanted are defined as matched at 12/12 HLA-alleles. We will include up to 7/8 (HLA-A, B, C, and DRB1) matched unrelated donors.
   3. One haplotype-mismatched related donors will be included.

Recipient Exclusion Criteria:

1. Pulmonary dysfunction defined as DLCO (corrected for hemoglobin and alveolar volume) < 35% of predicted OR baseline oxygen saturation of <85% or oxygen pressure in arterial blood (PaO2) <70.
2. Severe cardiac dysfunction defined as ejection fraction <45% or subjects who have been receiving chronic transfusion therapy for > 1 year and have evidence of iron overload (serum ferritin levels >1000 ng/mL), a cardiac MRI is required. Cardiac T2* <10 ms results in exclusion.
3. Liver iron content (LIC) ≥15 mg Fe/g dry weight on R2 MRI of liver, unless liver biopsy within 3 months prior to or at screening shows no evidence of bridging fibrosis or cirrhosis. Presence of bridging (portal to portal) fibrosis or cirrhosis in liver biopsy OR transaminases >5x normal upper limit (ULN) for age or direct bilirubin >3x normal upper limit (ULN).
4. Clinical stroke within 6 months of anticipated transplant
5. Karnofsky performance score < 50%
6. HIV infection
7. Uncontrolled viral, bacterial, fungal, or protozoal infection at the time of study enrollment.
8. Patient with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate HSCT in the opinion of the investigator.
9. Patient unable to understand the nature and risks inherent in the HSCT process.
10. History of non-compliance severe enough in the estimation of the treating team to preclude the patient from undergoing unrelated donor transplantation.
11. Patient is pregnant or lactating.
12. Inability to provide adequate transfusion support or increased risk immunohematological complications due presence of anti-RBC antibody against stem cell donor.
13. Presence of donor-specific HLA antibodies

Donor Eligibility and Selection Criteria

Please note, donor selection will follow our institutional standard operating procedure (SOP). Key criteria are summarized below for convenience:

1. Donor should be evaluated for eligibility to donate by an independent physician not directly caring for the patient on study protocol
2. Donor is willing to sign informed consent allowing the use of the peripheral blood stem cell (PBSC) product for the hematopoietic stem cell transplant (HSCT) of the recipient
3. Donor must meet HLA match criteria outlined in the inclusion criteria above
4. Donor cannot be pregnant or lactating and must agree to contraception until after the donation procedure is complete
5. Testing negative for HIV and viral hepatitis
6. Free of Hb S (defined as Hb S less than 50%) and other hemoglobinopathies that are symptomatic or of clinical significance
7. Targeted minimum stem cell dose of 5.0 x 10e6 CD34 cells/Kg (a marker of human hematopoietic stem cells) of recipient weight 8. Fulfills standard criteria for eligibility as a donor for hematopoietic stem cell transplant (HSCT)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Failure Rate | 12 Months Post Stem Cell Transplant
  Failure rate is a safety endpoint. Failure rate is defined as: graft failure (Primary Graft Rejection: Primary graft rejection is defined as the absence of donor cells (% donor cells < 5%) assessed by bone marrow or peripheral blood chimerism assays by Day 42. Late Graft Rejection: The absence (<5%) of donor hematopoietic cells in peripheral blood or bone marrow beyond Day 42 in a patient who had initial evidence of hematopoietic recovery with > 20% donor cells will be considered a late graft rejection.); or grades III-IV GVHD (as assessed by Center for International Blood and Marrow Transplant Research (CIBMTR) and NIH Consensus Criteria); or death at 100 days.

SECONDARY OUTCOMES:
Time to Engraftment | Day 100
  Time to neutrophil engraftment is defined as the first of 3 measurements on consecutive days when the patient has an absolute neutrophil count of 500/μL after conditioning. Time to platelet engraftment will be defined as the first day of a minimum of 3 measurements on different days that the patient has achieved a platelet count > 50,000/μL AND did not receive a platelet transfusion in the previous 7 days. Time to red cell engraftment is defined as the first of two measurements on different days that the patient has achieved an absolute reticulocyte count > 30,000/μL following conditioning regimen induced nadir.
Incidence of GVHD of Any Grade | 12 Months Post Stem Cell Transplant
  Incidence of acute and chronic GVHD of any grade as evaluated according to the CIBMTR and NIH criteria respectively.
Incidence of other transplant related toxicities | 12 Months Post Stem Cell Transplant
  Incidence of other transplant related toxicities, including Veno-occlusive disease (VOD), Idiopathic pneumonia syndrome (IPS), Central nervous system (CNS) toxicity, or Posterior reversible encephalopathy syndrome (PRES).
Incidence of Significant transplant-related infections | 12 Months Post Stem Cell Transplant
  Significant infections will be recorded including but not limited to bacterial or fungal sepsis, cytomegalovirus (CMV) reactivation with/without clinical disease, adenovirus infection, epstein-barr virus (EBV) reactivation with or without post-transplant lymphoproliferative disorders (PTLD), other significant viral reactivations or community-acquired viral infections and invasive mold infections.
Number of participants with donor chimerism >5% | Day 30, Day 100, and 1 year
  Chimerism is a measure of the engraftment of donor cells within the recipient and is expressed as the percentage ratio between the number of donor cells and recipient cells. Chimerism will be determined by Short Tandem Repeat analysis.
Percentage of Participants who Achieve Immune Reconstitution | 12 Months Post Stem Cell Transplant
  Peripheral blood quantitative assessment of the main lymphocyte subpopulations (CD3+, CD4+, CD8+, CD19+, and CD16+/56+). Lymphocytes will be assessed by flow cytometry. In addition, quantitative immunoglobulins will be measured for Immunoglobulin A (IgA), Immunoglobulin M (IgM) and Immunoglobulin (IgG). These will be performed at Day +60 (±10 days) as well as at 1 year (+/- 2 weeks) and after long term follow up at the discretion of the investigator. Descriptive statistics will be used to describe the percentage of patient who are able to achieve reconstitution of important lymphocyte subsets and B cell function at the defined timepoint above.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Y Mapara, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States